CLINICAL TRIAL: NCT03285295
Title: Abbott Laboratories Alinity s Blood Screening Assays - Clinical Evaluation Protocol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Diagnostics Division (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 9DY-02-14U01-03
Record Dates: First submitted 2017-09-12; First posted 2017-09-18 (Actual); Results first posted 2019-10-09 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-09

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Evaluation of assay performance characteristics.
  Participants:
  * Alinity s HBsAg: 17987
  * Alinity s HTLV I/II: 17685
  * Alinity s Anti-HCV: 17904
  * Alinity s HIV Ag/Ab Combo: 19571
  * Alinity s Anti-HBc: 16776
  * Alinity s Chagas: 16958
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Screening (Experimental): All subjects will be tested with at least one of the investigational Alinity s assays (Anti-HBc, Anti-HCV, HTLV I/II, Chagas, HBsAg, HBsAg Confirmatory, HIV Ag/Ab Combo) on Alinity s system.
  Interventions: Device: Alinity s HBsAg and Alinity s HBsAg Confirmatory Assay; Device: Alinity s HTLV I/II Assay; Device: Alinity s Anti-HCV Assay; Device: Alinity s HIV Ag/Ab Combo Assay; Device: Alinity s Anti-HBc Assay; Device: Alinity s Chagas Assay

INTERVENTIONS:
Device: Alinity s HBsAg and Alinity s HBsAg Confirmatory Assay — For all donor specimens with investigational Alinity s HBsAg and Alinity s HBsAg Confirmatory results that are discordant with final status after supplemental testing, an attempt will be made to obtain a follow-up whole blood specimen approximately 4 to 6 weeks after initial donation for further analysis.
Device: Alinity s HTLV I/II Assay — For all donor specimens with investigational Alinity s HTLV I/II results that are discordant with final status after supplemental testing, an attempt will be made to obtain a follow-up whole blood specimen approximately 4 to 6 weeks after initial donation for further analysis.
Device: Alinity s Anti-HCV Assay — For all donor specimens with investigational Alinity s Anti-HCV results that are discordant with final status after supplemental testing, an attempt will be made to obtain a follow-up whole blood specimen approximately 4 to 6 weeks after initial donation for further analysis.
Device: Alinity s HIV Ag/Ab Combo Assay — For all donor specimens with investigational Alinity s HIV Ag/Ab Combo results that are discordant with final status after supplemental testing, an attempt will be made to obtain a follow-up whole blood specimen approximately 4 to 6 weeks after initial donation for further analysis.
Device: Alinity s Anti-HBc Assay — For all donor specimens with investigational Alinity s Anti-HBc results that are discordant with final status after supplemental testing, an attempt will be made to obtain a follow-up whole blood specimen approximately 4 to 6 weeks after initial donation for further analysis.
Device: Alinity s Chagas Assay — For all donor specimens with investigational Alinity s Chagas results that are discordant with final status after supplemental testing, an attempt will be made to obtain a follow-up whole blood specimen approximately 4 to 6 weeks after initial donation for further analysis.

SUMMARY:
The objective of this study is to demonstrate the performance and intended use of each of the Alinity s investigational assays in a donor screening environment using clinical specimens to evaluate assay performance characteristics. A comparison of assay performance will be done versus the Food and Drug Administration (FDA) licensed assays. The data will be used to support regulatory submissions and/or publications.

DETAILED DESCRIPTION:
This study evaluates Alinity s investigational assays using the Alinity s System. The Alinity s System is a high-volume, automated, blood-screening analyzer that is designed to determine the presence of specific antigens and antibodies by using chemiluminescent microparticle immunoassay (CMIA) detection technology. The system performs high-throughput routine and stat processing that features continuous access and automated retesting.

The Alinity s System is used for infectious disease marker testing in blood-screening and plasma laboratories for the following assays: Anti-HBc, Anti-HCV, HTLV I/II, Chagas, HBsAg, HBsAg Confirmatory and HIV Ag/Ab Combo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy donors who consented to participate in the study.

Exclusion Criteria:

* For testing with the Alinity s Chagas assay, exclude donors that have been screened on a previous donation using a licensed test for antibodies to T cruzi.

Note: A subject may participate at different times during the study for separate assay studies, but each subject should be represented only once for each assay.

The protocol does not define an age limit. A donor must be at least 17 years old to donate to the general blood supply, or 16 years old with parental/guardian consent, if allowed by state law.

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 106881 (Actual)
Dates: Start 2017-09-15 (Actual); Primary Completion 2018-05-23 (Actual); Study Completion 2018-06-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy R Haley, M.D., Principal Investigator — Bloodworks Northwest; Thomas S Jones, Ph.D., Principal Investigator — QualTex Laboratories; Susan S Ganz, M.D., Principal Investigator — Biotest Pharmaceuticals Corporation; Toby L Simon, M.D., Principal Investigator — CSL Plasma Inc.; Susan L Stramer, Ph.D., Principal Investigator — American Red Cross National Testing Laboratory
Locations (5):
- United States (5):
  - Biotest Pharmaceuticals Corporation, Boca Raton, Florida
  - American Red Cross National Testing Laboratory, St Louis, Missouri
  - CSL Plasma Inc., Knoxville, Tennessee
  - QualTex Laboratories, San Antonio, Texas
  - Bloodworks Northwest, Renton, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Alinity s HBsAg: 17987 Alinity s HTLV I/II: 17685 Alinity s Anti-HCV: 17904 Alinity s HIV Ag/Ab Combo: 19571 Alinity s Anti-HBc: 16776 Alinity s Chagas: 16958
Groups:
- Specificity: US blood and/or plasmapheresis donor specimens collected as part of routine blood and/or plasma donation were tested with the investigational Alinity s HBsAg and HBsAg Confirmatory, HTLV I/II, Anti-HCV, HIV Ag/Ab Combo, Anti-HBc, and Chagas assays.
- Sensitivity: Specimens characterized as positive obtained from specimen vendors or collected under separate specimen collection protocols were tested by the investigational Alinity s HBsAg and HBsAg Confirmatory, HTLV I/II, Anti-HCV, HIV Ag/Ab Combo, Anti-HBc, and Chagas assays.
- Increased Risk Population: Specimens with Increased Risk of Infection obtained from specimen vendors or collected under separate specimen collection protocols were tested with investigational Alinity s assays. This population includes specimens from US population with risk for HBV, HTLV I/II, HCV, and HIV infection.
- Endemic Population: Specimens from endemic areas obtained from specimen vendors or collected under separate specimen collection protocols were tested with investigational Alinity s assays. This population includes specimens from individuals which reside in an HTLV I/II, HIV, and Chagas endemic area.
- HBV Recovered Population: Specimens classified as recovered HBV Infection based on 4 marker hepatitis testing obtained from specimen vendors or collected under separate specimen collection protocols were tested with investigational Alinity s HBsAg assay.
Period: Alinity s HBsAg
Arm/Group | Specificity | Sensitivity | Increased Risk Population | Endemic Population | HBV Recovered Population
Started | 17095 | 438 | 403 | 0 | 51
Completed | 16993 | 432 | 403 | 0 | 51
Not Completed | 102 | 6 | 0 | 0 | 0
Not completed — Protocol Violation | 11 | 0 | 0 | 0 | 0
Not completed — No Result on Comparator Assay | 17 | 0 | 0 | 0 | 0
Not completed — No Results Generated | 74 | 6 | 0 | 0 | 0
Period: Alinity s HBsAg Confirmatory
Arm/Group | Specificity | Sensitivity | Increased Risk Population | Endemic Population | HBV Recovered Population
Started | 8 | 432 | 3 | 0 | 0
Completed | 8 | 432 | 3 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Alinity s HBsAg Follow-Up
Arm/Group | Specificity | Sensitivity | Increased Risk Population | Endemic Population | HBV Recovered Population
Started | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Alinity s HTLV I/II
Arm/Group | Specificity | Sensitivity | Increased Risk Population | Endemic Population | HBV Recovered Population
Started | 15968 | 706 | 502 | 509 | 0
Completed | 15877 | 706 | 502 | 509 | 0
Not Completed | 91 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 6 | 0 | 0 | 0 | 0
Not completed — No Result on Comparator Assay | 15 | 0 | 0 | 0 | 0
Not completed — No Results Generated | 70 | 0 | 0 | 0 | 0
Period: Alinity s HTLV I/II Follow-Up
Arm/Group | Specificity | Sensitivity | Increased Risk Population | Endemic Population | HBV Recovered Population
Started | 12 | 0 | 0 | 0 | 0
Completed | 8 | 0 | 0 | 0 | 0
Not Completed | 4 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 4 | 0 | 0 | 0 | 0
Period: Alinity s Anti-HCV
Arm/Group | Specificity | Sensitivity | Increased Risk Population | Endemic Population | HBV Recovered Population
Started | 17095 | 402 | 407 | 0 | 0
Completed | 16999 | 402 | 407 | 0 | 0
Not Completed | 96 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 12 | 0 | 0 | 0 | 0
Not completed — No Results on Comparator Assay | 13 | 0 | 0 | 0 | 0
Not completed — No Results Generated | 71 | 0 | 0 | 0 | 0
Period: Alinity s Anti-HCV Follow-Up
Arm/Group | Specificity | Sensitivity | Increased Risk Population | Endemic Population | HBV Recovered Population
Started | 20 | 0 | 0 | 0 | 0
Completed | 2 | 0 | 0 | 0 | 0
Not Completed | 18 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 18 | 0 | 0 | 0 | 0
Period: Alinity s HIV Ag/Ab Combo
Arm/Group | Specificity | Sensitivity | Increased Risk Population | Endemic Population | HBV Recovered Population
Started | 17095 | 1336 | 605 | 535 (Individuals at Increased Risk of HIV Infection from HIV-2 Endemic Areas) | 0
Completed | 16996 | 1336 | 605 | 535 (Individuals at Increased Risk of HIV Infection from HIV-2 Endemic Areas) | 0
Not Completed | 99 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 11 | 0 | 0 | 0 | 0
Not completed — No Results on Comparator Assay | 16 | 0 | 0 | 0 | 0
Not completed — No Results Generated | 72 | 0 | 0 | 0 | 0
Period: Alinity s HIV Ag/Ab Combo Follow-Up
Arm/Group | Specificity | Sensitivity | Increased Risk Population | Endemic Population | HBV Recovered Population
Started | 15 | 0 | 0 | 0 | 0
Completed | 4 | 0 | 0 | 0 | 0
Not Completed | 11 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 11 | 0 | 0 | 0 | 0
Period: Alinity s Anti-HBc
Arm/Group | Specificity | Sensitivity | Increased Risk Population | Endemic Population | HBV Recovered Population
Started | 15968 | 405 | 403 | 0 | 0
Completed | 15877 | 404 | 403 | 0 | 0
Not Completed | 91 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 8 | 0 | 0 | 0 | 0
Not completed — No Results on Comparator Assay | 13 | 1 | 0 | 0 | 0
Not completed — No Results Generated | 70 | 0 | 0 | 0 | 0
Period: Alinity s Anti-HBc Follow-Up
Arm/Group | Specificity | Sensitivity | Increased Risk Population | Endemic Population | HBV Recovered Population
Started | 16 | 0 | 0 | 0 | 0
Completed | 2 | 0 | 0 | 0 | 0
Not Completed | 14 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 14 | 0 | 0 | 0 | 0
Period: Alinity s Chagas
Arm/Group | Specificity | Sensitivity | Increased Risk Population | Endemic Population | HBV Recovered Population
Started | 16023 | 320 | 0 | 615 | 0
Completed | 15804 | 320 | 0 | 615 | 0
Not Completed | 219 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 76 | 0 | 0 | 0 | 0
Not completed — No Results on Comparator Assay | 38 | 0 | 0 | 0 | 0
Not completed — No Results Generated | 105 | 0 | 0 | 0 | 0
Period: Alinity s Chagas Follow-Up
Arm/Group | Specificity | Sensitivity | Increased Risk Population | Endemic Population | HBV Recovered Population
Started | 14 | 0 | 0 | 0 | 0
Completed | 1 | 0 | 0 | 0 | 0
Not Completed | 13 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 13 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Donors and pedigree
Groups:
- Endemic Population: Specimens from endemic areas obtained from specimen vendors or collected under separate specimen collection protocols were tested with investigational Alinity s assays. This population includes specimens from individuals which reside in an HTLV I/II, HIV, and Chagas endemic areas.
- Total: Total of all reporting groups
Arm/Group | Specificity | Sensitivity | Increased Risk Population | Endemic Population | HBV Recovered Population | Total
Number analyzed (Participants) | 98546 | 3600 | 2320 | 1659 | 51 | 106176
Age, Customized [Count of Participants; unit: Participants]
  ≥16 years: Alinity s HBsAg | 16993 | 432 | 403 | 0 | 51 | 17879
  ≥16 years: Alinity s HTLV I/II | 15877 | 706 | 502 | 509 | 0 | 17594
  ≥16 years: Alinity s Anti-HCV | 16999 | 402 | 407 | 0 | 0 | 17808
  ≥16 years: Alinity s HIV Ag/Ab Combo | 16996 | 1336 | 605 | 535 | 0 | 19472
  ≥16 years: Alinity s Anti-HBc | 15877 | 404 | 403 | 0 | 0 | 16684
  ≥16 years: Alinity s Chagas | 15804 | 320 | 0 | 615 | 0 | 16739
Sex/Gender, Customized [Count of Participants; unit: Participants] — Population: Each row represents a different population as a subset of a total enrollment.
  Participants
    Alinity s HBsAg Gender: number analyzed (Participants) | 16993 | 432 | 403 | 0 | 51 | 17879
    Alinity s HBsAg Gender: Male | 0 | 312 | 288 | 0 | 23 | 623
    Alinity s HBsAg Gender: Female | 0 | 92 | 115 | 0 | 28 | 235
    Alinity s HBsAg Gender: Unknown | 16993 | 28 | 0 | 0 | 0 | 17021
    Alinity s HTLV I/II Gender: number analyzed (Participants) | 15877 | 706 | 502 | 509 | 0 | 17594
    Alinity s HTLV I/II Gender: Male | 0 | 182 | 335 | 316 | 0 | 833
    Alinity s HTLV I/II Gender: Female | 0 | 290 | 167 | 193 | 0 | 650
    Alinity s HTLV I/II Gender: Unknown | 15877 | 234 | 0 | 0 | 0 | 16111
    Alinity s Anti-HCV Gender: number analyzed (Participants) | 16999 | 402 | 407 | 0 | 0 | 17808
    Alinity s Anti-HCV Gender: Male | 0 | 241 | 291 | 0 | 0 | 532
    Alinity s Anti-HCV Gender: Female | 0 | 161 | 116 | 0 | 0 | 277
    Alinity s Anti-HCV Gender: Unknown | 16999 | 0 | 0 | 0 | 0 | 16999
    Alinity s HIV Ag/Ab Combo Gender: number analyzed (Participants) | 16996 | 1336 | 605 | 535 | 0 | 19472
    Alinity s HIV Ag/Ab Combo Gender: Male | 0 | 891 | 420 | 279 | 0 | 1590
    Alinity s HIV Ag/Ab Combo Gender: Female | 0 | 222 | 185 | 256 | 0 | 663
    Alinity s HIV Ag/Ab Combo Gender: Unknown | 16996 | 223 | 0 | 0 | 0 | 17219
    Alinity s Anti-HBc Gender: number analyzed (Participants) | 15877 | 404 | 403 | 0 | 0 | 16684
    Alinity s Anti-HBc Gender: Male | 0 | 230 | 288 | 0 | 0 | 518
    Alinity s Anti-HBc Gender: Female | 0 | 165 | 115 | 0 | 0 | 280
    Alinity s Anti-HBc Gender: Unknown | 15877 | 9 | 0 | 0 | 0 | 15886
    Alinity s Chagas Gender: number analyzed (Participants) | 15804 | 320 | 0 | 615 | 0 | 16739
    Alinity s Chagas Gender: Male | 0 | 104 | 0 | 216 | 0 | 320
    Alinity s Chagas Gender: Female | 0 | 102 | 0 | 399 | 0 | 501
    Alinity s Chagas Gender: Unknown | 15804 | 114 | 0 | 0 | 0 | 15918
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Each row represents a different population as a subset of a total enrollment.
  Participants
    Alinity s HBsAg Race/Ethnicity: number analyzed (Participants) | 16993 | 432 | 403 | 0 | 51 | 17879
    Alinity s HBsAg Race/Ethnicity: Asian | 0 | 24 | 3 | 0 | 1 | 28
    Alinity s HBsAg Race/Ethnicity: Black or African American | 0 | 123 | 244 | 0 | 6 | 373
    Alinity s HBsAg Race/Ethnicity: White | 0 | 45 | 79 | 0 | 13 | 137
    Alinity s HBsAg Race/Ethnicity: Hispanic or Latino | 0 | 33 | 71 | 0 | 2 | 106
    Alinity s HBsAg Race/Ethnicity: American Indian or Alaskan Native | 0 | 0 | 3 | 0 | 0 | 3
    Alinity s HBsAg Race/Ethnicity: Other | 0 | 23 | 3 | 0 | 2 | 28
    Alinity s HBsAg Race/Ethnicity: Unknown | 16993 | 184 | 0 | 0 | 27 | 17204
    Alinity s HTLV I/II Race/Ethnicity: number analyzed (Participants) | 15877 | 706 | 502 | 509 | 0 | 17594
    Alinity s HTLV I/II Race/Ethnicity: Asian | 0 | 26 | 4 | 0 | 0 | 30
    Alinity s HTLV I/II Race/Ethnicity: Black or African American | 0 | 63 | 154 | 305 | 0 | 522
    Alinity s HTLV I/II Race/Ethnicity: White | 0 | 114 | 256 | 0 | 0 | 370
    Alinity s HTLV I/II Race/Ethnicity: Hispanic or Latino | 0 | 224 | 87 | 204 | 0 | 515
    Alinity s HTLV I/II Race/Ethnicity: American Indian or Alaskan Native | 0 | 5 | 1 | 0 | 0 | 6
    Alinity s HTLV I/II Race/Ethnicity: Other | 0 | 7 | 0 | 0 | 0 | 7
    Alinity s HTLV I/II Race/Ethnicity: Unknown | 15877 | 267 | 0 | 0 | 0 | 16144
    Alinity s Anti-HCV Race/Ethnicity: number analyzed (Participants) | 16999 | 402 | 407 | 0 | 0 | 17808
    Alinity s Anti-HCV Race/Ethnicity: Asian | 0 | 0 | 2 | 0 | 0 | 2
    Alinity s Anti-HCV Race/Ethnicity: Black or African American | 0 | 95 | 239 | 0 | 0 | 334
    Alinity s Anti-HCV Race/Ethnicity: White | 0 | 14 | 100 | 0 | 0 | 114
    Alinity s Anti-HCV Race/Ethnicity: Hispanic or Latino | 0 | 12 | 62 | 0 | 0 | 74
    Alinity s Anti-HCV Race/Ethnicity: American Indian or Alaskan Native | 0 | 0 | 1 | 0 | 0 | 1
    Alinity s Anti-HCV Race/Ethnicity: Other | 0 | 0 | 1 | 0 | 0 | 1
    Alinity s Anti-HCV Race/Ethnicity: Unknown | 16999 | 281 | 2 | 0 | 0 | 17282
    Alinity s HIV Ag/Ab Combo Race/Ethnicity: number analyzed (Participants) | 16996 | 1336 | 605 | 535 | 0 | 19472
    Alinity s HIV Ag/Ab Combo Race/Ethnicity: Asian | 0 | 4 | 5 | 0 | 0 | 9
    Alinity s HIV Ag/Ab Combo Race/Ethnicity: Black or African American | 0 | 364 | 404 | 535 | 0 | 1303
    Alinity s HIV Ag/Ab Combo Race/Ethnicity: White | 0 | 286 | 115 | 0 | 0 | 401
    Alinity s HIV Ag/Ab Combo Race/Ethnicity: Hispanic or Latino | 0 | 430 | 81 | 0 | 0 | 511
    Alinity s HIV Ag/Ab Combo Race/Ethnicity: American Indian or Alaskan Native | 0 | 5 | 0 | 0 | 0 | 5
    Alinity s HIV Ag/Ab Combo Race/Ethnicity: Other | 0 | 4 | 0 | 0 | 0 | 4
    Alinity s HIV Ag/Ab Combo Race/Ethnicity: Unknown | 16996 | 243 | 0 | 0 | 0 | 17239
    Alinity s Anti-HBc Race/Ethnicity: number analyzed (Participants) | 15877 | 404 | 403 | 0 | 0 | 16684
    Alinity s Anti-HBc Race/Ethnicity: Asian | 0 | 5 | 3 | 0 | 0 | 8
    Alinity s Anti-HBc Race/Ethnicity: Black or African American | 0 | 40 | 244 | 0 | 0 | 284
    Alinity s Anti-HBc Race/Ethnicity: White | 0 | 39 | 79 | 0 | 0 | 118
    Alinity s Anti-HBc Race/Ethnicity: Hispanic or Latino | 0 | 4 | 71 | 0 | 0 | 75
    Alinity s Anti-HBc Race/Ethnicity: American Indian or Alaskan Native | 0 | 1 | 3 | 0 | 0 | 4
    Alinity s Anti-HBc Race/Ethnicity: Other | 0 | 18 | 3 | 0 | 0 | 21
    Alinity s Anti-HBc Race/Ethnicity: Unknown | 15877 | 297 | 0 | 0 | 0 | 16174
    Alinity s Chagas Race/Ethnicity: number analyzed (Participants) | 15804 | 320 | 0 | 615 | 0 | 16739
    Alinity s Chagas Race/Ethnicity: Asian | 0 | 0 | 0 | 0 | 0 | 0
    Alinity s Chagas Race/Ethnicity: Black or African American | 0 | 0 | 0 | 0 | 0 | 0
    Alinity s Chagas Race/Ethnicity: White | 0 | 1 | 0 | 9 | 0 | 10
    Alinity s Chagas Race/Ethnicity: Hispanic or Latino | 0 | 205 | 0 | 576 | 0 | 781
    Alinity s Chagas Race/Ethnicity: American Indian or Alaskan Native | 0 | 0 | 0 | 30 | 0 | 30
    Alinity s Chagas Race/Ethnicity: Other | 0 | 0 | 0 | 0 | 0 | 0
    Alinity s Chagas Race/Ethnicity: Unknown | 15804 | 114 | 0 | 0 | 0 | 15918
Region of Enrollment [Count of Participants; unit: Participants] — Population: Each row represents a different country with populations within that country as a subset of a total enrollment for each assay.
  Not collected represents total number across all Alinity s assays: HBsAg, HTLV I/II, Anti-HCV, HIV Ag/Ab Combo, Anti-HBc, and Chagas.
  Participants
    United States: number analyzed (Participants) | 98546 | 3394 | 2320 | 0 | 51 | 104311
    United States: Alinity s HBsAg | 16993 | 0 | 403 | 0 | 0 | 17396
    United States: Alinity s HTLV I/II | 15877 | 0 | 0 | 0 | 0 | 15877
    United States: Alinity s Anti-HCV | 16999 | 0 | 407 | 0 | 0 | 17406
    United States: Alinity s HIV Ag/Ab Combo | 16996 | 0 | 605 | 0 | 0 | 17601
    United States: Alinity s Anti-HBc | 15877 | 0 | 403 | 0 | 0 | 16280
    United States: Alinity s Chagas | 15804 | 114 | 0 | 0 | 0 | 15918
    United States: Not collected | 0 | 3280 | 502 | 0 | 51 | 3833
    Haiti: number analyzed (Participants) | 0 | 0 | 0 | 204 | 0 | 204
    Haiti: Alinity s HBsAg | 0 | 0 | 0 | 0 | 0 | 0
    Haiti: Alinity s HTLV I/II | 0 | 0 | 0 | 204 | 0 | 204
    Haiti: Alinity s Anti-HCV | 0 | 0 | 0 | 0 | 0 | 0
    Haiti: Alinity s HIV Ag/Ab Combo | 0 | 0 | 0 | 0 | 0 | 0
    Haiti: Alinity s Anti-HBc | 0 | 0 | 0 | 0 | 0 | 0
    Haiti: Alinity s Chagas | 0 | 0 | 0 | 0 | 0 | 0
    Haiti: Not collected | 0 | 0 | 0 | 0 | 0 | 0
    Africa: number analyzed (Participants) | 0 | 0 | 0 | 635 | 0 | 635
    Africa: Alinity s HBsAg | 0 | 0 | 0 | 0 | 0 | 0
    Africa: Alinity s HTLV I/II | 0 | 0 | 0 | 100 | 0 | 100
    Africa: Alinity s Anti-HCV | 0 | 0 | 0 | 0 | 0 | 0
    Africa: Alinity s HIV Ag/Ab Combo | 0 | 0 | 0 | 535 | 0 | 535
    Africa: Alinity s Anti-HBc | 0 | 0 | 0 | 0 | 0 | 0
    Africa: Alinity s Chagas | 0 | 0 | 0 | 0 | 0 | 0
    Africa: Not collected | 0 | 0 | 0 | 0 | 0 | 0
    Mexico: number analyzed (Participants) | 0 | 9 | 0 | 100 | 0 | 109
    Mexico: Alinity s HBsAg | 0 | 0 | 0 | 0 | 0 | 0
    Mexico: Alinity s HTLV I/II | 0 | 0 | 0 | 0 | 0 | 0
    Mexico: Alinity s Anti-HCV | 0 | 0 | 0 | 0 | 0 | 0
    Mexico: Alinity s HIV Ag/Ab Combo | 0 | 0 | 0 | 0 | 0 | 0
    Mexico: Alinity s Anti-HBc | 0 | 0 | 0 | 0 | 0 | 0
    Mexico: Alinity s Chagas | 0 | 9 | 0 | 100 | 0 | 109
    Mexico: Not collected | 0 | 0 | 0 | 0 | 0 | 0
    South America: number analyzed (Participants) | 0 | 197 | 0 | 521 | 0 | 718
    South America: Alinity s HBsAg | 0 | 0 | 0 | 0 | 0 | 0
    South America: Alinity s HTLV I/II | 0 | 0 | 0 | 205 | 0 | 205
    South America: Alinity s Anti-HCV | 0 | 0 | 0 | 0 | 0 | 0
    South America: Alinity s HIV Ag/Ab Combo | 0 | 0 | 0 | 0 | 0 | 0
    South America: Alinity s Anti-HBc | 0 | 0 | 0 | 0 | 0 | 0
    South America: Alinity s Chagas | 0 | 197 | 0 | 316 | 0 | 513
    South America: Not collected | 0 | 0 | 0 | 0 | 0 | 0
    Central America: number analyzed (Participants) | 0 | 0 | 0 | 199 | 0 | 199
    Central America: Alinity s HBsAg | 0 | 0 | 0 | 0 | 0 | 0
    Central America: Alinity s HTLV I/II | 0 | 0 | 0 | 0 | 0 | 0
    Central America: Alinity s Anti-HCV | 0 | 0 | 0 | 0 | 0 | 0
    Central America: Alinity s HIV Ag/Ab Combo | 0 | 0 | 0 | 0 | 0 | 0
    Central America: Alinity s Anti-HBc | 0 | 0 | 0 | 0 | 0 | 0
    Central America: Alinity s Chagas | 0 | 0 | 0 | 199 | 0 | 199
    Central America: Not collected | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Alinity s HBsAg Assay Specificity
Description: Total of 16993 serum and plasma specimens from whole blood donors as well as plasmapheresis specimens were tested with Alinity s HBsAg Assay. Repeatedly reactive specimens were further tested with Alinity s HBsAg Confirmatory and supplemental assays, if required.
Time Frame: 10 months
Population: All blood and plasmapheresis donor specimens tested with Alinity s HBsAg assay per protocol.
Measure: Count of Participants; unit: Participants
Groups:
- Alinity s HBsAg Assay Specificity: US blood and plasmapheresis donor specimens collected as part of routine blood and plasma donation were tested with the investigational Alinity s assay.
Arm/Group | Alinity s HBsAg Assay Specificity
Number analyzed (Participants) | 16993
Participants
  Alinity s HBsAg Nonreactive HBsAg Negative | 16985
  Alinity s HBsAg Repeatedly Reactive HBsAg Negative | 6
  Alinity s HBsAg Positive | 2
Statistical Analysis 1: Comparison: Alinity s HBsAg Assay Specificity; Test type: Superiority; Binomial Distribution; Specificity sample size is a minimum of 15,000 donors; Clinical Specificity (%) = 99.96, 95% CI 2-sided [99.92 to 99.99]

2. Primary Outcome: Alinity s HBsAg and HBsAg Confirmatory Assay Sensitivity
Description: Total of 432 specimens from subjects known to be HBsAg positive were tested with Alinity s HBsAg and HBsAg Confirmatory assay.
Time Frame: 10 months
Population: Specimens from 432 individuals known to be positive for HBsAg were tested with Alinity s HBsAg and HBsAg Confirmatory assay per protocol.
Measure: Count of Participants; unit: Participants
Groups:
- Alinity s HBsAg and HBsAg Confirmatory Assay Sensitivity: Preselected HBsAg positive samples were obtained from specimen vendors or collected under separate specimen collection protocols were tested by the investigational Alinity s HBsAg and HBsAg Confirmatory assays. This population included individuals with acute hepatitis B infection, and individuals with chronic hepatitis B infection. HBV classification was determined using 4 HBV reference marker testing or medically diagnosed.
Arm/Group | Alinity s HBsAg and HBsAg Confirmatory Assay Sensitivity
Number analyzed (Participants) | 432
Participants
  Alinity s HBsAg Nonreactive | 0
  Alinity s HBsAg Reactive Confirmed | 432
  Alinity s HBsAg Reactive Not Confirmed | 0
Statistical Analysis 1: Comparison: Alinity s HBsAg and HBsAg Confirmatory Assay Sensitivity; Test type: Other — 95% Confidence Interval provided; Sensitivity; Point Estimate = 100.00, 95% CI 2-sided [99.15 to 100.00]

3. Primary Outcome: Alinity s HTLV I/II Assay Specificity
Description: Total of 15877 serum and plasma specimens from whole blood donors specimens were tested with Alinity s HTLV I/II Assay. Repeatedly reactive specimens were further tested with Alinity s HTLV I/II and supplemental assays, if required.
Time Frame: 10 months
Population: All blood donor specimens tested with Alinity s HTLV I/II assay per protocol.
Measure: Count of Participants; unit: Participants
Groups:
- Alinity s HTLV I/II Assay Specificity: US blood donor specimens collected as part of routine blood and plasma donation were tested with the investigational Alinity s HTLV I/II assay.
Arm/Group | Alinity s HTLV I/II Assay Specificity
Number analyzed (Participants) | 15877
Participants
  Alinity s HTLV Nonreactive HTLV Neg | 15864
  Alinity s HTLV Repeatedly Reactive HTLV Neg | 2
  HTLV Positive or Indeterminate | 11
Statistical Analysis 1: Comparison: Alinity s HTLV I/II Assay Specificity; Test type: Superiority; Binomial Distribution; Clinical Specificity (%) = 99.99, 95% CI 2-sided [99.95 to 100.00]

4. Primary Outcome: Alinity s HTLV I/II Assay Sensitivity
Description: Total of 706 specimens from subjects known to be HTLV positive were tested with Alinity s HTLV I/II assay. The population consists of the following:
  Anti-HTLV I Positive n = 461 Anti-HTLV II positive n = 141 Anti-HTLV III positive - Undifferentiated n = 4 Individual with HTLV I/II Associated Diseases n = 100
Time Frame: 10 months
Population: Specimens from 706 individuals known to be positive for HTLV were tested with Alinity s HTLV I/II assay per protocol.
Measure: Count of Participants; unit: Participants
Groups:
- Alinity s HTLV I/II Assay Sensitivity: This population includes both archived and leftover not individually identifiable specimens that are extensively characterized. The specimens were confirmed positive by research use only HTLV-I Western blot and HTLV-I and HTLV-II radioimmunoprecipitation assay (RIPA) and typed as HTLV-I or HTLV-II by immunofluorescence assay (IFA) titration.
  Individuals with HTLV-I/II Associated Diseases includes specimens prospectively collected from individuals diagnosed with adult T-cell leukemia/lymphoma (ATL) or HTLV-I associated myelopathy/tropical spastic paraparesis (HAM/TSP) using IRB-approved protocols sponsored by specimen vendors.
Arm/Group | Alinity s HTLV I/II Assay Sensitivity
Number analyzed (Participants) | 706
Participants
  Alinity s HTLV I/II Nonreactive | 0
  Alinity s HTLV I/II Repeatedly Reactive | 706
Statistical Analysis 1: Comparison: Alinity s HTLV I/II Assay Sensitivity; Test type: Other — 95% Confidence Interval provided; Sensitivity; Point Estimate = 100.00, 95% CI 2-sided [99.48 to 100.00]

5. Primary Outcome: Alinity s Anti-HCV Assay Specificity
Description: Total of 16,999 serum and plasma specimens from whole blood donors as well as plasmapheresis specimens were tested with Alinity s Anti-HCV assay. Repeatedly reactive specimens were tested further with supplemental assays, if required.
Time Frame: 10 months
Population: All blood and plasmapheresis donor specimens tested with Alinity s Anti-HCV assay per protocol.
Measure: Count of Participants; unit: Participants
Groups:
- Alinity s Anti-HCV Assay Specificity: US blood and plasmapheresis donor specimens collected as part of routine blood and plasma donation were tested with the investigational Alinity s Anti-HCV assay.
Arm/Group | Alinity s Anti-HCV Assay Specificity
Number analyzed (Participants) | 16999
Participants
  Alinity s Anti-HCV Nonreactive HCV Negative | 16975
  Alinity s Anti-HCV Repeatedly Reactive HCV Neg | 14
  HCV Positive or Indeterminate | 10
Statistical Analysis 1: Comparison: Alinity s Anti-HCV Assay Specificity; Test type: Superiority; Binomial Distribution; Clinical Specificity (%) = 99.92, 95% CI 2-sided [99.86 to 99.95]

6. Primary Outcome: Alinity s Anti-HCV Assay Sensitivity
Description: Total of 402 specimens from subjects known to be Anti-HCV positive were tested with Alinity s Anti-HCV assay.
Time Frame: 10 months
Population: Specimens from 402 individuals known to be positive for Anti-HCV were tested with Alinity s Anti-HCV assay per protocol.
Measure: Count of Participants; unit: Participants
Groups:
- Alinity s Anti-HCV Assay Sensitivity: This population includes specimens prospectively collected using IRB-approved protocols sponsored by Abbott Laboratories and vendor-collected leftover specimens that were not individually identifiable. A subset of these specimens was confirmed positive by an HCV recombinant immunoblot assay (RIBA). The remaining specimens were collected from subjects with a medical diagnosis of chronic HCV infection and history of greater than 6 months of HCV RNA/anti-HCV positivity. For these specimens, a current anti-HCV result was obtained.
Arm/Group | Alinity s Anti-HCV Assay Sensitivity
Number analyzed (Participants) | 402
Participants
  Alinity s Anti-HCV Nonreactive | 0
  Alinity s Anti-HCV Repeatedly Reactive | 402
Statistical Analysis 1: Comparison: Alinity s Anti-HCV Assay Sensitivity; Test type: Other — 95% Confidence Interval provided; Sensitivity; Point Estimate = 100.00, 95% CI 2-sided [99.09 to 100.00]

7. Primary Outcome: Alinity s HIV Ag/Ab Combo Assay Specificity
Description: Total of 16996 serum and plasma specimens from whole blood donors as well as plasmapheresis specimens were tested with Alinity s HIV Ag/Ab Combo Assay. Repeatedly reactive specimens were further tested with supplemental assays, if required.
Time Frame: 10 months
Population: All fresh whole blood and plasmapheresis donor specimens tested with Alinity s HIV Ag/Ab Combo assay per protocol.
Measure: Count of Participants; unit: Participants
Groups:
- Alinity s HIV Ag/Ab Combo Assay Specificity: US blood and plasmapheresis donor specimens collected as part of routine blood and plasma donation were tested with the investigational Alinity s HIV Ag/Ab Combo assay.
Arm/Group | Alinity s HIV Ag/Ab Combo Assay Specificity
Number analyzed (Participants) | 16996
Participants
  Alinity s HIV Nonreactive HIV Negative | 16981
  Alinity s HIV Repeatedly Reactive HIV Negative | 13
  HIV Indeterminate | 2
Statistical Analysis 1: Comparison: Alinity s HIV Ag/Ab Combo Assay Specificity; Test type: Superiority; Binomial Exact; Clinical Specificity (%) = 99.92, 95% CI 2-sided [99.87 to 99.96]

8. Primary Outcome: Alinity s HIV Ag/Ab Combo Assay Sensitivity
Description: Total of 1336 specimens from subjects known to be HIV-1/2 positive were tested with Alinity s HIV Ag/Ab Combo assay.
Time Frame: 10 months
Population: Specimens from 1336 individuals known to be positive for HIV-1/2 were tested with Alinity s HIV Ag/Ab Combo assay per protocol.
Measure: Count of Participants; unit: Participants
Groups:
- Alinity s HIV Ag/Ab Combo Assay Sensitivity: Preselected HIV-1/2 positive samples were obtained from specimen vendors or collected under separate specimen collection protocols were tested by the investigational Alinity s HIV Ag/Ab Combo assays. This population included individuals with HIV-1 and HIV-2 infection. The HIV-1 specimens were confirmed positive by HIV-1 Western blot and categorized by revised surveillance case definitions for HIV infection (2008) as stage 1 (n=488), stage 2 (n=427) or stage 3 (n=101) using CD4 counts and associated diagnosis. The specimens were confirmed positive for HIV-2 by HIV-2 Western blot and typed as HIV-2 only by Bio-Rad Multispot HIV-1/HIV-2 Rapid Test.The remaining are for Anti-HIV 2 (n=232), HIV-1 antigen (n=35), and HIV-1 viral isolates (n=53).
Arm/Group | Alinity s HIV Ag/Ab Combo Assay Sensitivity
Number analyzed (Participants) | 1336
Participants
  Alinity s HIV Ag/Ab Combo Nonreactive | 0
  Alinity s HIV Ag/Ab Combo Repeatedly Reactive Pos | 1336
  Alinity s HIV Ag/Ab Combo Repeatedly Reactive Neg | 0
Statistical Analysis 1: Comparison: Alinity s HIV Ag/Ab Combo Assay Sensitivity; Test type: Other — 95% Confidence Interval provided; Sensitivity; Point Estimate = 100.00, 95% CI 2-sided [99.72 to 100.00]

9. Primary Outcome: Alinity s Anti-HBc Assay Specificity
Description: Total of 15877 serum and plasma specimens from whole blood donor specimens were tested with Alinity s Anti-HBc Assay. Repeatedly reactive specimens were further tested with supplemental assays, if required.
Time Frame: 10 months
Population: All fresh whole blood donor specimens tested with Alinity s Anti-HBc assay per protocol.
Measure: Count of Participants; unit: Participants
Groups:
- Alinity s Anti-HBc Assay Specificity: US blood donor specimens collected as part of routine blood and plasma donation were tested with the investigational Alinity s Anti-HBc assay.
Arm/Group | Alinity s Anti-HBc Assay Specificity
Number analyzed (Participants) | 15877
Participants
  Alinity s Anti-HBc Nonreactive Anti-HBc Negative | 15833
  Alinity s Anti-HBc Repeatedly Reactive AntiHBc Neg | 16
  Anti-HBc Positive | 28
Statistical Analysis 1: Comparison: Alinity s Anti-HBc Assay Specificity; Test type: Superiority; Binomial Exact; Clinical Specificity (%) = 99.90, 95% CI 2-sided [99.84 to 99.94]

10. Primary Outcome: Alinity s Anti-HBc Assay Sensitivity
Description: Total of 404 specimens from individuals with hepatitis B infection were tested with investigational Alinity s Anti-HBc assay. The population consists of the following:
  Acute Hepatitis B infection n = 28 Chronic Hepatitis B infection n = 97 Recovered Hepatitis B infection n = 279
Time Frame: 10 months
Population: Specimens from 404 individuals with Hepatitis B infection were tested with Alinity s Anti-HBc assay per protocol.
Measure: Count of Participants; unit: Participants
Groups:
- Alinity s Anti-HBc Assay Sensitivity: Preselected Anti-HBc Positive specimens were obtained from individuals with acute hepatitis B infection, individuals with chronic hepatitis B infection, and individuals with recovered hepatitis B infection.
Arm/Group | Alinity s Anti-HBc Assay Sensitivity
Number analyzed (Participants) | 404
Participants
  Alinity s Anti-HBc Nonreactive | 0
  Alinity s Anti-HBc Repeatedly Reactive Positive | 404
  Alinity s Anti-HBc Repeatedly Reactive Negative | 0
Statistical Analysis 1: Comparison: Alinity s Anti-HBc Assay Sensitivity; Test type: Other — 95% Confidence Interval provided; Sensitivity; Point Estimate = 100.00, 95% CI 2-sided [99.09 to 100.00]

11. Primary Outcome: Alinity s Chagas Assay Specificity
Description: Total of 15804 serum and plasma specimens from whole blood donors specimens were tested with Alinity s Chagas Assay. Repeatedly reactive specimens were further tested with Alinity s Chagas and supplemental assays, if required.
Time Frame: 10 months
Population: All blood donor specimens tested with Alinity s Chagas assay per protocol.
Measure: Count of Participants; unit: Participants
Groups:
- Alinity s Chagas Assay Specificity: US blood donor specimens collected as part of routine blood and plasma donation were tested with the investigational Alinity s Chagas assay.
Arm/Group | Alinity s Chagas Assay Specificity
Number analyzed (Participants) | 15804
Participants
  Alinity s Chagas Nonreactive Chagas Negative | 15787
  Alinity s Chagas Repeatedly Reactive Chagas Neg | 3
  Chagas Positive or Indeterminate | 14
Statistical Analysis 1: Comparison: Alinity s Chagas Assay Specificity; Test type: Superiority; Binomial Exact; Clinical Specificity (%) = 99.98, 95% CI 2-sided [99.94 to 100.00]

12. Primary Outcome: Alinity s Chagas Assay Sensitivity
Description: Total of 320 specimens from subjects known to be Chagas positive were tested with investigational Alinity s Chagas assay.
Time Frame: 10 months
Population: Specimens from 320 individuals known to be positive for Chagas were tested with investigational Alinity s Chagas assay per protocol.
Measure: Count of Participants; unit: Participants
Groups:
- Alinity s Chagas Assay Sensitivity: Preselected T cruzi Parasitology Positive (n = 112) and preselected T cruzi Serology Positive (n = 208) samples were obtained from specimen vendors or collected under separate specimen collection protocols were tested by the investigational Alinity s Chagas assay.
Arm/Group | Alinity s Chagas Assay Sensitivity
Number analyzed (Participants) | 320
Participants
  Alinity s Chagas Nonreactive | 0
  Alinity s Chagas Repeatedly Reactive Positive | 320
  Alinity s Chagas Repeatedly Reactive Negative | 0
Statistical Analysis 1: Comparison: Alinity s Chagas Assay Sensitivity; Test type: Other — 95% Confidence Interval provided; Sensitivity; Point Estimate = 100.00, 95% CI 2-sided [98.85 to 100.00]

13. Secondary Outcome: Alinity s HBsAg Assay Increased Risk of HBV Infection
Description: Total of 403 specimens from subjects known to be at increased risk for HBV infection were tested with investigational Alinity s HBsAg assay.
  Sensitivity and Specificity not applicable.
Time Frame: 10 months
Population: Specimens from 403 individuals with increased risk for HBV infection were tested with Alinity s HBsAg assay per protocol.
Measure: Count of Participants; unit: Participants
Groups:
- Alinity s HBsAg Assay Increased Risk of HBV Infection: Specimens with Increased Risk of Infection obtained from specimen vendors or collected under separate specimen collection protocols were tested with investigational Alinity s assays. This population includes specimens from US population with risk for HBV infection.
Arm/Group | Alinity s HBsAg Assay Increased Risk of HBV Infection
Number analyzed (Participants) | 403
Participants
  Alinity s HBsAg Nonreactive Negative | 400
  Alinity s HBsAg Nonreactive Positive | 0
  Alinity s HBsAg Reactive Confirmed | 3
  Alinity s HBsAg Reactive Not Confirmed | 0

14. Secondary Outcome: Alinity s HBsAg Assay Recovered HBV Infection
Description: Total of 51 specimens from subjects classified as recovered HBV infection were tested with investigational Alinity s HBsAg assay.
  Sensitivity/Specificity calculation for this population not applicable.
Time Frame: 10 months
Population: Specimens from 51 individuals classified as recovered HBV infection were tested with Alinity s HBsAg assay per protocol.
Measure: Count of Participants; unit: Participants
Groups:
- Alinity s HBsAg Assay Recovered HBV Infection: Specimens classified as recovered HBV Infection based on 4 marker hepatitis testing obtained from specimen vendors or collected under separate specimen collection protocols were tested with investigational Alinity s HBsAg assay.
Arm/Group | Alinity s HBsAg Assay Recovered HBV Infection
Number analyzed (Participants) | 51
Participants
  Alinity s HBsAg Nonreactive Negative | 51
  Alinity s HBsAg Nonreactive Positive | 0
  Alinity s HBsAg Reactive Confirmed | 0
  Alinity s HBsAg Reactive Not Confirmed | 0

15. Secondary Outcome: Alinity s HTLV Assay Increased Risk of HTLV Infection
Description: Total of 502 specimens from subjects known to be at increased risk for HTLV I/II infection were tested with investigational Alinity s HTLV I/II assay.
  Sensitivity and Specificity not applicable.
Time Frame: 10 months
Population: Specimens from 502 individuals with increased risk for HTLV I/II infection were tested with Alinity s HTLV I/II assay per protocol.
Measure: Count of Participants; unit: Participants
Groups:
- Alinity s HTLV Assay Increased Risk of HTLV-I/II Infection: Specimens with Increased Risk of Infection obtained from specimen vendors or collected under separate specimen collection protocols were tested with investigational Alinity s assays. This population includes specimens from US population with risk for HTLV I/II infection.
Arm/Group | Alinity s HTLV Assay Increased Risk of HTLV-I/II Infection
Number analyzed (Participants) | 502
Participants
  Alinity s HTLV I/II Nonreactive Negative | 491
  Alinity s HTLV I/II Nonreactive Positive | 0
  Alinity s HTLV I/II Nonreactive Indeterminate | 0
  Alinity s HTLV I/II Reactive Indeterminate | 0
  Alinity s HTLV I/II Reactive Positive | 11
  Alinity s HTLV I/II Reactive Negative | 0

16. Secondary Outcome: Alinity s HTLV I/II Assay Endemics
Description: Total of 509 specimens from subjects collected from areas known to be endemic for HTLV I/II infection were tested with investigational Alinity s HTLV I/II assay. Sensitivity and Specificity not applicable.
Time Frame: 10 months
Population: Specimens from 509 individuals collected from areas known to be endemic for HTLV I/II infection were tested with Alinity s HTLV I/II assay per protocol.
Measure: Count of Participants; unit: Participants
Groups:
- Alinity s HTLV I/II Assay Endemics: Specimens from endemic areas obtained from specimen vendors or collected under separate specimen collection protocols were tested with investigational Alinity s assays. This population includes specimens from individuals which reside in an HTLV I/II endemic area.
Arm/Group | Alinity s HTLV I/II Assay Endemics
Number analyzed (Participants) | 509
Participants
  Alinity s HTLV I/II Nonreactive Negative | 495
  Alinity s HTLV I/II Nonreactive Positive | 0
  Alinity s HTLV I/II Nonreactive Indeterminate | 4
  Alinity s HTLV I/II Reactive Indeterminate | 0
  Alinity s HTLV I/II Reactive Positive | 10
  Alinity s HTLV I/II Reactive Negative | 0

17. Secondary Outcome: Alinity s Anti-HCV Assay Increased Risk for HCV
Description: Total of 407 specimens from subjects known to be at increased risk for HCV infection were tested with investigational Alinity s Anti-HCV assay.
Time Frame: 10 months
Population: Specimens from 407 individuals with increased risk for HCV infection were tested with Alinity s Anti-HCV assay per protocol.
Measure: Count of Participants; unit: Participants
Groups:
- Alinity s Anti-HCV Assay Increased Risk for HCV: Specimens with Increased Risk of Infection obtained from specimen vendors or collected under separate specimen collection protocols were tested with investigational Alinity s assays. This population includes specimens from US population with risk for HCV infection.
Arm/Group | Alinity s Anti-HCV Assay Increased Risk for HCV
Number analyzed (Participants) | 407
Participants
  Alinity s Anti-HCV Nonreactive Negative | 316
  Alinity s Anti-HCV Noreactive Positive | 0
  Alinity s Anti-HCV Nonreactive Indeterminate | 0
  Alinity s Anti-HCV Reactive Indeterminate | 0
  Alinity s Anti-HCV Reactive Positive | 90
  Alinity s Anti-HCV Reactive Negative | 1
Statistical Analysis 1: Comparison: Alinity s Anti-HCV Assay Increased Risk for HCV; Sensitivity; Test type: Other — 95% Confidence Interval provided; Sensitivity; Point Estimate = 100.00, 95% CI 2-sided [95.98 to 100.00]

18. Secondary Outcome: Alinity s HIV Ag/Ab Combo Assay Increased Risk of HIV-1/2
Description: Total of 605 specimens from subjects known to be at increased risk for HIV-1/2 infection were tested with investigational Alinity s HIV Ag/Ab Combo assay.
  Sensitivity and Specificity not applicable.
Time Frame: 10 months
Population: Specimens from 605 individuals with increased risk for HIV-I/2 infection were tested with Alinity s HIV Ag/Ab Combo assay per protocol.
Measure: Count of Participants; unit: Participants
Groups:
- Alinity s HIV Ag/Ab Combo Assay Increased Risk for HIV-1/2: Specimens with Increased Risk of Infection obtained from specimen vendors or collected under separate specimen collection protocols were tested with investigational Alinity s assays. This population includes specimens from US population with risk for HIV infection.
Arm/Group | Alinity s HIV Ag/Ab Combo Assay Increased Risk for HIV-1/2
Number analyzed (Participants) | 605
Participants
  Alinity s HIV Ag/Ab Combo Nonreactive Negative | 582
  Alinity s HIV Ag/Ab Combo Nonreactive Positive | 0
  Alinity s HIV Ag/Ab Comb Nonreactive Indeterminate | 0
  Alinity s HIV Ag/Ab Combo Reactive Indeterminate | 0
  Alinity s HIV Ag/Ab Combo Reactive Positive | 21
  Alinity s HIV Ag/Ab Combo Reactive Negative | 2

19. Secondary Outcome: Alinity s HIV Ag/Ab Combo Assay Endemics
Description: Total of 535 specimens from subjects collected from areas known to be endemic for HIV infection were tested with investigational Alinity s HIV Ag/Ab Combo assay.
Time Frame: 10 months
Population: Specimens from 535 individuals collected from areas known to be endemic for HIV infection were tested with Alinity s HIV Ag/Ab Combo assay per protocol.
Measure: Count of Participants; unit: Participants
Groups:
- Alinity s HIV Ag/Ab Combo Assay Endemics: Specimens from endemic areas obtained from specimen vendors or collected under separate specimen collection protocols were tested with investigational Alinity s assays. This population includes specimens from individuals which reside in an HIV endemic area.
Arm/Group | Alinity s HIV Ag/Ab Combo Assay Endemics
Number analyzed (Participants) | 535
Participants
  Alinity s HIV Ag/Ab Combo Nonreactive Negative | 472
  Alinity s HIV Ag/Ab Combo Nonreactive Positive | 0
  Alinity s HIV Ag/Ab Comb Nonreactive Indeterminate | 2
  Alinity s HIV Ag/Ab Combo Reactive Indeterminate | 10
  Alinity s HIV Ag/Ab Combo Reactive Positive | 49
  Alinity s HIV Ag/Ab Combo Reactive Negative | 2
Statistical Analysis 1: Comparison: Alinity s HIV Ag/Ab Combo Assay Endemics; Sensitivity; Test type: Other — 95% Confidence Interval provided; Sensitivity; Point Estimate = 100.00, 95% CI 2-sided [92.75 to 100.00]

20. Secondary Outcome: Alinity s Anti-HBc Assay Increased Risk for HBV
Description: Total of 403 specimens from subjects known to be at increased risk for HBV infection were tested with investigational Alinity s Anti-HBc assay.
Time Frame: 10 months
Population: Specimens from 403 individuals with increased risk for HBV infection were tested with Alinity s Anti-HBc assay per protocol.
Measure: Count of Participants; unit: Participants
Groups:
- Alinity s Anti-HBc Assay Increased Risk for HBV: Specimens with Increased Risk of Infection obtained from specimen vendors or collected under separate specimen collection protocols were tested with investigational Alinity s assays. This population includes specimens from US population with risk for HBV infection
Arm/Group | Alinity s Anti-HBc Assay Increased Risk for HBV
Number analyzed (Participants) | 403
Participants
  Alinity s Anti-HBc Nonreactive Negative | 319
  Alinity s Anti-HBc Nonreactive Positive | 0
  Alinity s Anti-HBc Reactive Positive | 70
  Alinity s Anti-HBc Reactive Negative | 14
Statistical Analysis 1: Comparison: Alinity s Anti-HBc Assay Increased Risk for HBV; Sensitivity; Test type: Other — 95% Confidence Interval provided; Sensitivity; Point Estimate = 100.00, 95% CI 2-sided [94.87 to 100.00]

21. Secondary Outcome: Alinity s Chagas Assay Endemics
Description: Total of 615 specimens from subjects collected from areas known to be endemic for Chagas infection were tested with investigational Alinity s Chagas assay
Time Frame: 10 months
Population: Specimens from 615 subjects collected from areas known to be endemic for Chagas infection were tested with Alinity s Chagas assay per protocol.
Measure: Count of Participants; unit: Participants
Groups:
- Alinity s Chagas Assay Endemics: Specimens from endemic areas obtained from specimen vendors or collected under separate specimen collection protocols were tested with investigational Alinity s assays. This population includes specimens from individuals which reside in Chagas endemic area.
Arm/Group | Alinity s Chagas Assay Endemics
Number analyzed (Participants) | 615
Participants
  Alinity s Chagas Nonreactive Negative | 466
  Alinity s Chagas Noreactive Positive | 2
  Alinity s Chagas Nonreactive Indeterminate | 0
  Alinity s Chagas Reactive Indeterminate | 0
  Alinity s Chagas Reactive Positive | 146
  Alinity s Chagas Reactive Negative | 1
Statistical Analysis 1: Comparison: Alinity s Chagas Assay Endemics; Sensitivity; Test type: Other — 95% Confidence Interval provided; Sensitivity; Point Estimate = 98.65, 95% CI 2-sided [95.20 to 99.84]

ADVERSE EVENTS:
Time Frame: Subject adverse events related to blood collection during the 3-6 months of donor follow-up specimen collection.
Description: Subject adverse event reporting was only applicable to donors that returned for follow-up specimen collection.
  Adverse events were not applicable for blood and plasmapheresis donor specimens collected as part of routine blood donation and specimens provided by Abbott to testing sites.
  There were no subject or device adverse events associated with testing.
Groups:
- Alinity s HBsAg Follow-Up Specimen Collection: For all donor specimens with investigational Alinity s results that are discordant with final status after supplemental testing, an attempt will be made to obtain a follow-up whole blood specimen approximately 4 to 6 weeks after initial donation for further analysis.
  No donors required for follow-up collection for Alinity s HBsAg study.
- Alinity s HTLV I/II Follow-Up Specimen Collection: For all donor specimens with investigational Alinity s results that are discordant with final status after supplemental testing, an attempt will be made to obtain a follow-up whole blood specimen approximately 4 to 6 weeks after initial donation for further analysis.
  12 donors were eligible for follow-up collection for Alinity s HTLV I/II study. 8 out of 12 were able to provide follow-up specimen.
- Alinity s Anti-HCV Follow-Up Specimen Collection: For all donor specimens with investigational Alinity s results that are discordant with final status after supplemental testing, an attempt will be made to obtain a follow-up whole blood specimen approximately 4 to 6 weeks after initial donation for further analysis.
  20 donors were eligible for follow-up collection for Alinity s Anti-HCV study. 2 out of 20 were able to provide follow-up specimen.
- Alinity s HIV Ag/Ab Combo Follow-Up Specimen Collection: For all donor specimens with investigational Alinity s results that are discordant with final status after supplemental testing, an attempt will be made to obtain a follow-up whole blood specimen approximately 4 to 6 weeks after initial donation for further analysis.
  15 donors were eligible for follow-up collection for Alinity s HIV Ag/Ab Combo study.
  4 out of 15 were able to provide follow-up specimen.
- Alinity s Anti-HBc Follow-Up Specimen Collection: For all donor specimens with investigational Alinity s results that are discordant with final status after supplemental testing, an attempt will be made to obtain a follow-up whole blood specimen approximately 4 to 6 weeks after initial donation for further analysis.
  16 donors were eligible for follow-up collection for Alinity s Anti-HBc study. 2 out of 16 were able to provide follow-up specimen.
- Alinity s Chagas Follow-Up Specimen Collection: For all donor specimens with investigational Alinity s results that are discordant with final status after supplemental testing, an attempt will be made to obtain a follow-up whole blood specimen approximately 4 to 6 weeks after initial donation for further analysis.
  14 donors were eligible for follow-up collection for Alinity s Chagas study.
  1 out of 14 were able to provide follow-up specimen.
Arm/Group | Alinity s HBsAg Follow-Up Specimen Collection | Alinity s HTLV I/II Follow-Up Specimen Collection | Alinity s Anti-HCV Follow-Up Specimen Collection | Alinity s HIV Ag/Ab Combo Follow-Up Specimen Collection | Alinity s Anti-HBc Follow-Up Specimen Collection | Alinity s Chagas Follow-Up Specimen Collection
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/8 | 0/2 | 0/4 | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/8 | 0/2 | 0/4 | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/8 | 0/2 | 0/4 | 0/2 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI must provide a copy of any proposed publication/presentation at least 60 days prior to submission for sponsor's review/approval. The PI must incorporate changes as the sponsor requires in order to protect the sponsor's proprietary rights and interests. The sponsor may require the PI to include acknowledgement of the sponsor's role in the study. The PI may be requested to delay publication/presentation an extra 60 days to enable sponsor to secure patent or other proprietary protection.

DOCUMENTS (5):
  • Informed Consent Form: Alinity s Follow-Up Study - Donor Consent for Central IRB (2017-08-17): https://cdn.clinicaltrials.gov/large-docs/95/NCT03285295/ICF_000.pdf
  • Informed Consent Form: Alinity s Follow-Up Study - Donor Consent for Local IRB (2017-11-17): https://cdn.clinicaltrials.gov/large-docs/95/NCT03285295/ICF_001.pdf
  • Study Protocol and Statistical Analysis Plan (2018-04-24): https://cdn.clinicaltrials.gov/large-docs/95/NCT03285295/Prot_SAP_002.pdf
  • Informed Consent Form: Information Sheet for Central IRB (2017-08-23): https://cdn.clinicaltrials.gov/large-docs/95/NCT03285295/ICF_003.pdf
  • Informed Consent Form: Information Sheet for Local IRB (2017-11-17): https://cdn.clinicaltrials.gov/large-docs/95/NCT03285295/ICF_004.pdf